CLINICAL TRIAL: NCT04592614
Title: Choose to Move: How Can Health Benefits of an Effective, Scaled-up, Health Promotion Model for Older Adults be Sustained?
Brief Title: Choose to Move - Next Steps: Can 'Booster Sessions' Sustain Health Benefits of an Effective, Scaled-up, Health Promotion Program?
Acronym: CTM-NS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Active Aging Society (Other)
Responsible Party: Principal Investigator, Heather McKay, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GR012151; PJT-169159 (Other Grant/Funding Number: Canadian Institutes of Health Research); H20-00780 (Other: University of British Columbia)
Record Dates: First submitted 2020-09-22; First posted 2020-10-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Aging; Mobility Limitation; Sedentary Behavior; Loneliness; Social Isolation
Keywords: Physical Inactivity; Sustainability; Maintenance; Behaviour Change; Physical Activity; Implementation Science; Scale-up
MeSH Terms: conditions — Mobility Limitation; Sedentary Behavior; Social Isolation; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment intervention model.
  Consenting participants (older adults and activity coaches) will be randomly assigned (at the level of their CTM group) to one of two CTM-NS study arms: 1) monthly virtual group meetings (high dose), or 2) quarterly virtual group meetings (low dose). Randomization is not relevant for provincial partners and coordinators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (Experimental): CTM-NS participants receiving monthly virtual group meetings for 2 years (24 meetings total)
  Interventions: Behavioral: Choose to Move - Next Steps
- Low dose (Experimental): CTM-NS participants receiving quarterly virtual group meetings for 2 years (8 meetings total)
  Interventions: Behavioral: Choose to Move - Next Steps

INTERVENTIONS:
Behavioral: Choose to Move - Next Steps — Choose to Move - Next Steps consists of a series of group meetings delivered virtually for 2 years. Group meetings (1-hr each) of 6-11 older adults will be facilitated by a trained Activity Coach and delivered remotely via the Zoom or GoToMeeting platform (password protected; access through phone or internet). Each group meeting will provide information on a health-related topic of interest and will include time for goal setting, discussion and sharing among participants. Older adults will have the option to sign up for a bi-weekly CTM electronic newsletter containing health information and ideas and resources for older adults to be physically active and socially connected at home (and elsewhere as local restrictions permit). Activity Coaches will also facilitate social connections between participants to encourage contact (by phone or online) outside of group sessions (for interested participants only).

SUMMARY:
One-third of Canadians will be older adults (>65y) by 2050. Thus, healthy aging is a public health priority. Many older adult health promoting interventions have been implemented, yet few were scaled-up and sustained. Choose to Move (CTM) is an effective, adaptable, community-based health promotion program for older adults. CTM, co-created with government and community stakeholders, has been scaled-up across British Columbia (BC) using a phased approach (2015-2021). The investigators evaluated the impact of CTM on the health of seniors who participated and the results were extremely positive: CTM increased mobility, physical activity, social connectedness and improved mental health indicators like loneliness. When these outcomes were assessed again, one year after the end of CTM, these improvements had diminished.

In this trial the investigators aim to determine if health benefits of CTM can be maintained by providing ongoing support to CTM participants. Booster interventions have been defined as "brief contacts beyond the main part of the intervention to reinforce previous intervention content" (Fjeldsoe et al., 2011, p. 601). Choose to Move - Next Steps (CTM-NS) is a two-year intervention where participants who recently completed CTM will receive different doses of a 'booster' program. Specifically, participants will be randomly allocated to virtual group meetings on a monthly (study arm 1; high dose) or quarterly (study arm 2; low dose) basis. Group meetings will be facilitated by an Activity Coach.

Objectives:

The investigators will conduct 1) impact, 2) implementation, and 3) economic evaluations of CTM-NS across 24 months.

Hypotheses:

For objective 1, the investigators hypothesize that improvements in older adult participant outcomes (primary outcome: mobility; secondary outcomes: physical activity, loneliness, social isolation, social connectedness, sitting time, screen time, social network, health status) obtained during CTM will be maintained over the 2 year CTM-NS study. Participants in the monthly group meetings (study arm 1) will maintain benefits to a greater degree than participants in the quarterly group meetings (study arm 2). Objectives 2 and 3 are descriptive and therefore have no hypotheses.

DETAILED DESCRIPTION:
Study Design

The investigators will use a type 2 hybrid effectiveness-implementation study design. CTM participants who choose to enrol in CTM-NS will be randomly assigned to one of two CTM-NS booster intervention arms: high dose (monthly meetings) or low dose (quarterly meetings).

Participants and Recruitment

There are 4 participant groups in this study:

1. Provincial partners. These are individuals who make strategic and policy decisions for their organization. Provincial partners will be invited to participate in the study through written invitation and consent form delivered via email from a member of the research team. These individuals will be asked to respond to the invite and confirm or decline participation.
2. Provincial coordinators. These individuals coordinate and oversee delivery of programs within delivery partner organizations. Provincial coordinators will be invited to participate in the study through written invitation and consent form delivered via email from a member of the research team. They will be asked to respond to the invite and confirm or decline participation.
3. Activity Coaches. Activity Coaches are hired and contracted by delivery partners to deliver CTM-NS. They will be informed of the evaluation and invited to participate during hiring and training.
4. Older adults. CTM evaluation participants who have recently completed CTM will be invited to participate in CTM-NS.

Intervention and Randomization

Participants will be randomized (along with any other participants from the same CTM group) by a member of the research team to one of two CTM-NS study arms. The sustainability portion of the intervention will be 24 months and consist of monthly (study arm 1; high dose) or quarterly (study arm 2; low dose) group meetings delivered remotely via the Zoom or GoToMeeting platform (password protected; access through phone or internet). Group meetings (1-hr each) of 6-11 older adults will be facilitated by a trained Activity Coach. Older adults will have the option to sign up for a bi-weekly CTM electronic newsletter containing health information and ideas and resources for older adults to be physically active and socially connected at home (and elsewhere as local restrictions permit). Within each group, Activity Coaches will also facilitate social connections between participants to encourage contact (by phone or online) outside of group sessions (for interested participants only). Groups will be combined as needed to achieve and maintain targeted group sizes. The CTM-NS intervention is only open to older adults who participated in the CTM evaluation.

Timeline

CTM will be delivered in 2 cycles:

1. CTM Fall 2020 cycle with program start dates approximately Sept-Oct 2020;
2. CTM Winter 2021 cycle with program start dates approximately Jan-Feb 2021.

Corresponding CTM-NS program start dates are approximately Jan-Feb 2021 (for Fall 2020 CTM programs) and April-May 2021 (for Winter 2021 CTM programs).

CTM-NS Evaluation

The investigators will use a type 2 hybrid effectiveness-implementation study design and mixed (qualitative and quantitative) methods to address the research objectives.

Participant groups will be evaluated as follows:

1. Provincial partners will be interviewed at 12 and 24 months after the start of the first CTM-NS program. In this group the investigators assess: adaptation; innovation characteristics; community context (facilitators and barriers to implementation; sustainability of delivery).
2. Provincial coordinators will be interviewed at 12 and 24 months after the start of the first CTM-NS program. In this group the investigators assess: reach; adaptation; community context (facilitators and barriers to implementation, sustainability of delivery); innovation characteristics; prevention support system; economic evaluation (costs associated with delivering CTM-NS).
3. Activity Coaches will provide survey data at 3, 12, and 24 months of each CTM-NS program they deliver. A subset of Activity Coaches (n=20) will be interviewed at 3, 12, and 24 months. In this group the investigators assess: dose delivered; quality; participant responsiveness; adaptation; provider characteristics; innovation characteristics; community context (facilitators and barriers to implementation); prevention support system.
4. Older adults will provide survey data at 0, 3, 12, and 24 months of their CTM-NS program. A subset of older adults (n=20) will be interviewed at 3, 12, and 24 months. In this group the investigators assess: reach (participant characteristics); dose received; participant responsiveness (satisfaction, engagement, enjoyment); quality; impact of CTM-NS on participant-level outcomes; how contextual factors influence program engagement and participant-level outcomes. Thus, participants will provide data at 4 time points in total: 0 (baseline for CTM-NS), 3, 12 and 24 months. Participants' baseline data from the main CTM study will be used in combination with these data to assess sustainability of outcomes (post-CTM is equivalent to baseline CTM-NS).

ELIGIBILITY:
Inclusion Criteria:

* Provincial partners inclusion criteria: These are individuals who make strategic and policy decisions for their organization
* Provincial coordinators inclusion criteria: These individuals coordinate and oversee delivery of programs within our delivery partner organizations.
* Activity Coach inclusion criteria: Completed CTM training and able to connect to the Zoom or GoToMeeting platform via internet (video and audio required in order to see and hear participants) for online programs
* Older adult inclusion criteria: English speaking, age ≥60 yrs, self-described as engaging in <150 min of moderate-to-vigorous physical activity per week and demonstrated readiness for physical activity (by the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+), Get Active Questionnaire or a letter of recommendation from their physician) before joining CTM, able to connect to the Zoom or GoToMeeting platform via phone or internet in order to participate in virtual group meetings (for online programs only), currently (or recently completed) participating in CTM evaluation

Exclusion Criteria:

* Provincial partners, provincial coordinators and Activity Coach exclusion criteria: None
* Older adult exclusion criteria: Non-English speaking, Unable to connect to the Zoom or GoToMeeting platform via phone or internet in order to participate in virtual group meetings

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 424 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change in mobility limitations | 0, 3, 12, 24 months
  Two items will assess change in a participants' ability to walk a quarter of a mile and up 10 steps (Simonsick et al., 2008). The output variable is self-reported presence of mobility-disability (no/any difficulty walking 400m or climbing one flight of stairs).
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in physical functioning | 0, 3, 12, 24 months
  Change in mobility will be assessed with the Physical Functioning Subscale of the 36-Item Short Form Survey (SF-36; Ware et al., 1989). The measure asks participants to rate if their health limits them in performing 10 different activities. The output variable is an average score from 0-100 of physical functioning, where a higher score indicates a more favourable health state.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in self-perception of mobility | 0, 3, 12, 24 months
  The Mobility Assessment Tool-Short Form (MAT-sf; Rejeski et al., 2015) will be used to assess change in mobility. The MAT-sf is a validated, short form video-animated tool to assess participant self-perception of mobility. Only participants with an internet connection are able to complete this measure. The output variable is a self-rated mobility score (30-80), with higher scores indicating greater self-perception of mobility.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.

SECONDARY OUTCOMES:
Change in physical activity | 0, 3, 12, 24 months
  The single item physical activity questionnaire will be used to measure change in physical activity (Milton, Bull & Bauman, 2011). Output variable is self-reported number of days/week ≥30 min PA in the past week.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in loneliness | 0, 3, 12, 24 months
  The three-item loneliness scale (Hughes et al., 2004) will be used to assess change in loneliness. Participants rate three aspects of loneliness. The output variable is loneliness score (3-9); lower scores indicate lower levels of loneliness.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in social isolation | 0, 3, 12, 24 months
  Change in social isolation will be assessed using a 4-item questionnaire adapted from Vernoff, Kulka & Douvan (1981). The output variable is social isolation score (0-15). Lower scores indicate greater levels of social isolation and higher scores indicate lower levels of social isolation.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in social connectedness | 0, 3, 12, 24 months
  A single item measure from the My Health My Community survey (2014) will be used to assess change in sense of belonging as an indicator of social connectedness. The output variable is sense of belonging score (1-4) with lower scores indicating a stronger sense of belonging.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in sitting time | 0, 3, 12, 24 months
  A five-item questionnaire (Marshall et al., 2010) will be used to assess change in sitting time (hours and minutes) each day in the following domains: (a) while travelling to and from places (e.g., work, shops); (b) while at work; (c) while watching television; (d) while using a computer at home; and (e) at leisure not including watching television (e.g., visiting friends, movies, eating out) on a weekday and a weekend day. The output variables are sitting hours per day across 5 domains.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in screen time | 0, 3, 12, 24 months
  A single item from the My Health My Community survey (My Health My Community, 2013) will be used to assess change in screen time. The output variable is the range of hours of screen time per day.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in social network | 0, 3, 12, 24 months
  Change in participant social network will be assessed using the 6-item Lubben Social Network Questionnaire (Lubben et al., 2006). The output variable is a social network score (range 0 to 30) where higher scores indicate larger social networks.
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in health status (EQ-5D-5L Profile) | 0, 3, 12, 24 months
  Change in health status (EQ-5D-5L Profile) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. Responses are used to create a 5-digit number which will be used descriptively.
  Change will be assessed descriptively across 0, 3, 12 and 24 months.
Change in health status (EQ-5D-5L Level Sum Score) | 0, 3, 12, 24 months
  Change in health status (EQ-5D-5L Level Sum Score) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. The Level Sum Score uses the 5-digit profile to create a numeric score, with scores ranging from 5-25 (lower levels indicate lower levels of perceived problems).
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.
Change in health status (EQ-5D-5L Visual Analogue Scale) | 0, 3, 12, 24 months
  Change in health status (EQ-5D-5L Visual Analogue Scale) will be assessed with the EQ-5D-5L (The EuroQol Group, 1990). Participants report on their health on a visual analogue scale from 0 (worst health) to 100 (best health).
  Change will be assessed using longitudinal modelling across 0, 3, 12 and 24 months.

OTHER OUTCOMES:
Reach - Individual | 24 months
  Reach is defined as the proportion of the intended priority audience who participate in the intervention (Saunders et al., 2005).
  Reach of CTM-NS will be captured across 3, 12 and 24 months at the level of the participant. This is operationalized as the number of older adult participants (and proportion of eligible population).
  Data will be provided by Provincial Coordinators (program records).
Reach - Organizational | 24 months
  Reach is defined as the proportion of the intended priority audience who participate in the intervention (Saunders et al., 2005).
  Reach of CTM-NS will be captured across 3, 12 and 24 months at the level of organizations. This is operationalized as the number of Activity Coaches and sites that deliver CTM-NS.
  Data will be provided by Provincial Coordinators (program records).
Dose delivered (Intervention Components) | 24 months
  Dose delivered is defined as the amount of each intervention component delivered or provided to participants (Saunders et al 2005). This will be captured at 3, 12, and 24 months.
  Dose delivered (by Activity Coaches) will be assessed via survey. Items have been designed in-house. For example, "I provided opportunities for group check-in with Choose to Move participants during virtual group meetings", with response options on a scale from 0-4 (no/a few/most/all group meetings).
Dose delivered (Implementation Strategies) | 24 months
  Dose delivered is defined as the amount of each implementation strategy delivered or provided to participants (Saunders et al 2005). This will be captured at 3, 12, and 24 months.
  Data will be collected from internal program records.
Dose received | 24 months
  Dose received is defined as the amount of each intervention component received by participants (attendance). This will be captured at 3, 12, and 24 months time points.
  Activity Coaches will provide dose received (by older adults) data via survey. Items have been designed in-house. For example, Activity Coaches will be asked "How many group meetings did this participant attend?". Attendance will be expressed as a percentage out of 24 (for participants in the high dose arm) and 8 (for participants in the low dose arm).
Quality | 24 months
  Defined as how well different program components were conducted (e.g., are the main program elements delivered clearly and correctly?) (Durlak and Dupre 2008) and the extent to which the intervention was implemented as planned (Saunders et al., 2005).
  The extent to which Activity Coaches deliver CTM-NS with quality will be captured at 3, 12, and 24 months. Older adults will provide data via survey. Items have been designed in-house and response options will be on an agreement scale or yes/no (e.g., "I feel comfortable at the Choose to Move group meetings.").
Participant responsiveness | 24 months
  Defined as the degree to which CTM-NS stimulates the interest or holds the attention of participants (Durlak and Dupre 2008).
  Older adult participant satisfaction, engagement and enjoyment with each component of CTM-NS will be captured at 3, 12, and 24 months. Data will be collected from Activity Coaches and older adults via survey. Items have been designed in-house (e.g., "Participants were enthusiastic, interested, and engaged with the CTM content and each other during virtual group meetings."), and response options will include agreement scales and yes/no.
Adaptation (survey) | 24 months
  Defined as changes made to the original program during implementation (Durlak and Dupre, 2008).
  Adaptation of CTM-NS during delivery will be described and characterized using an adaptation framework (Stirman et al 2019). Activity Coaches will provide data via survey across 3, 12, and 24 months. Items have been designed in-house and include open-ended responses. For example, "When you delivered Choose to Move to this group of participants, did you make any adaptations or modifications? These could be additions, deletions, substitutions, repetitions, etc. If so, please describe the modification(s), explain why you made them, and explain when and/or the frequency with which you made them."
  Open-ended responses will be explored using framework analysis.
Adaptation (interviews) | 24 months
  Defined as changes made to the original program during implementation (Durlak and Dupre, 2008).
  Data to be provided by Provincial coordinators (interview) and Activity Coaches (focus groups). Interview and focus group guides were designed in-house (e.g., "We described and outlined the structure of the Choose to Move program in your training supplement, but we acknowledge that it is not always feasible or realistic to deliver it as planned. Can you tell me about any changes you made to the program, if any?").
  Interview and focus group data will be explored using framework analysis.
Community context (survey) | 24 months
  Defined as aspects of the larger social, political, and economic environment that may influence intervention implementation (Linnan & Steckler, 2002).
  The context (policy, health, community) in which CTM-NS is delivered that may support and/or hinder program implementation will be captured at 3, 12, and 24 months. Data will be provided by Activity Coaches via survey.
  Items have been designed in-house (e.g., "What factors helped you to deliver Choose to Move?", with a list of response options).
Community context (interviews) | 24 months
  Defined as aspects of the larger social, political, and economic environment that may influence intervention implementation (Linnan & Steckler, 2002).
  Data will be provided by Provincial partners, Provincial coordinators (interviews) and Activity Coaches (focus groups). Interview guides have been designed in-house (e.g., "How does offering CTM fit with the strategic direction of your organization moving forward?").
  Interview and focus group data will be explored using framework analysis.
Provider characteristics (interviews) | 24 months
  Defined as aspects of the provider that may influence intervention implementation (e.g., organizational functioning).
  CTM-NS provider characteristics that support and/or hinder program implementation (perceived need, readiness, self-efficacy) will be captured at 3, 12, and 24 months. Data will be provided by Activity Coaches (focus groups) and Provincial coordinators (interviews). Interview scripts have been designed in-house (e.g. "Are there any major challenges your organization needs to overcome to continue to deliver CTM?").
  Interview and focus group data will be explored using framework analysis.
Innovation characteristics (Acceptability) | 24 months
  Innovation characteristics are defined as aspects of the intervention that may influence implementation. Acceptability is the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory (Proctor et al., 2011).
  Four items, each rated 1-5, will be used to assess acceptability of CTM-NS as perceived by Provincial Partners and Activity Coaches (Weiner et al., 2017) across at time points 3, 12, and 24 months via survey. The output variable is a mean score from 1-5, with higher scores indicating more acceptable.
Innovation characteristics (Feasibility) | 24 months
  Innovation characteristics are defined as aspects of the intervention that may influence implementation. Feasibility is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting (Proctor et al., 2011)
  Four items, each rated 1-5, will be used to assess feasibility of CTM-NS as perceived by Provincial Partners and Activity Coaches (Weiner et al., 2017) across at time points 3, 12, and 24 months via survey. The output variable is a mean score from 1-5, with higher scores indicating more feasible.
Innovation characteristics (Appropriateness) | 24 months
  Innovation characteristics are defined as aspects of the intervention that may influence implementation. Appropriateness is the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer; and/ or perceived fit of the innovation to address a particular issue or problem (Proctor et al 2011)
  Four items, each rated 1-5, will be used to assess appropriateness of CTM-NS as perceived by Provincial Partners and Activity Coaches (Weiner et al., 2017) across at time points 3, 12, and 24 months via survey. The output variable is a mean score from 1-5, with higher scores indicating more appropriate.
Innovation characteristics (survey) | 24 months
  Innovation characteristics are defined as aspects of the intervention that may influence implementation.
  Feasibility, acceptability and appropriateness of CTM-NS as perceived by older adults (Weiner et al., 2017) will be captured across at time points 3, 12, and 24 months via survey. Items have been designed in-house. For example, older adults will be asked, "Overall how easy is it for you to attend virtual group meetings?".
Innovation characteristics (interviews) | 24 months
  Defined as aspects of the intervention that may influence implementation.
  Data provided by Provincial Partners/Coordinators (interviews) and Activity Coaches (focus groups). Interview guides have been designed in-house. For example, Activity Coaches will be asked "What factors do you think helped with the delivery of the model? What worked well during program delivery?".
  Interview and focus group data will be explored using framework analysis.
Prevention support system (survey) | 24 months
  Defined as aspects of the support system that may influence implementation (e.g., training and technical assistance).
  Characteristics of the prevention support system that support and/or hinder program implementation (satisfaction with training and support) will be assessed. Activity Coaches will provide data via survey. Questions have been designed in-house (e.g., "The Choose to Move training provided me with the resources I needed to deliver CTM-NS."), and response options will include agreement scales and yes/no.
Prevention support system (interviews) | 24 months
  Defined as aspects of the support system that may influence implementation (e.g., training and technical assistance).
  Characteristics of the prevention support system that support and/or hinder program implementation (satisfaction with training and support) will be assessed. Data provided by Provincial Coordinators and Activity Coaches via interview/focus groups. Interview questions have been designed in-house (e.g., "What was the support like from the Active Aging Research Team throughout the planning and delivery phases of Choose to Move?").
  Interview and focus group data will be explored using framework analysis.
Direct intervention delivery costs | 24 months
  Direct intervention delivery costs (overall, per program and per participant) will be assessed at the end of CTM-NS.
  Data will be provided by Provincial Coordinators via project management records, including expenditures across all aspects of program development and implementation (e.g., program costs, personnel and non-personnel costs, recruitment, and organizational/equipment costs).
Value | 24 months
  Value will be assessed by comparing the incremental cost per participant with benefit achieved at the participant level across each study arm. It will be calculated at the end of the CTM-NS.
  Financial data proved by Provincial Coordinators via project management records.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A McKay, PhD, Principal Investigator — University of British Columbia; Joanie Sims-Gould, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Hip Health and Mobility, Robert H.N. Ho Research Centre, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Marshall AL, Miller YD, Burton NW, Brown WJ. Measuring total and domain-specific sitting: a study of reliability and validity. Med Sci Sports Exerc. 2010 Jun;42(6):1094-102. doi: 10.1249/MSS.0b013e3181c5ec18. PMID 19997030
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Simonsick EM, Newman AB, Visser M, Goodpaster B, Kritchevsky SB, Rubin S, Nevitt MC, Harris TB; Health, Aging and Body Composition Study. Mobility limitation in self-described well-functioning older adults: importance of endurance walk testing. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):841-7. doi: 10.1093/gerona/63.8.841. PMID 18772472
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. Health Promot Pract. 2005 Apr;6(2):134-47. doi: 10.1177/1524839904273387. PMID 15855283
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Wiltsey Stirman S, Baumann AA, Miller CJ. The FRAME: an expanded framework for reporting adaptations and modifications to evidence-based interventions. Implement Sci. 2019 Jun 6;14(1):58. doi: 10.1186/s13012-019-0898-y. PMID 31171014
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Fjeldsoe B, Neuhaus M, Winkler E, Eakin E. Systematic review of maintenance of behavior change following physical activity and dietary interventions. Health Psychol. 2011 Jan;30(1):99-109. doi: 10.1037/a0021974. PMID 21299298
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- See also: Website for the Choose to Move Program — http://www.choosetomove.ca/